CLINICAL TRIAL: NCT05964114
Title: Prospective Individualization of the First Vancomycin Dose Using Population Pharmacokinetic Models.
Brief Title: First Time Right of Vancomycin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Sebastiaan D.T. Sassen, PharmD PhD, Pharmacometrician, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7646
Record Dates: First submitted 2023-01-24; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Vancomycin; Pharmacokinetics
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Starting dose of vancomycin standard vs MIPD (Experimental): Comparison of vancomycin initial dosing via standard of care (flat dose adjusted for renal function) versus model informed precision dosing (starting dose adjusted using pharmacokinetic models).
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Initial dosing based on (a combinations of) pharmacokinetic models tailored to the individual patient. Dose adjustment starting dose (within registered dosing range).

SUMMARY:
In 2020, only 16% of the Intensive Care Unit (ICU) patients achieved therapeutic drug concentrations after continuous administration of the first vancomycin dose. Many beneficial population pharmacokinetic (PPK) models are available however these are prevented from being widely implemented in daily practice due to the complexity. The aim of this study is to evaluate the effectiveness of individualized dosing with PPK models using a newly developed user-friendly pharmacokinetic (PK) tool.

In a preceding retrospective study, the percentage of patients within the target range after initiation of continuous vancomycin increased from 28% to 39% (excluding CRRT and ECMO patients) with calculated concentrations based on theoretical dose adjustments. In this study we want to prospectively evaluate the concentration of vancomycin at 24, 28 and 72 hours after the start of treatment with individualized dosages based on (a combination) of available PPK models in 134 adult ICU and orthopedic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who receive continuous vancomycin treatment at the ICU or orthopaedic department
* Patient or their legal representative is able and willing to sign the Informed Consent Form

Exclusion Criteria:

* Pregnant woman
* Children
* Patients with a transplantation history
* Patients on continuous renal replacement therapy (CRRT)
* Patients receiving extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients within target range of vancomycin for standard treatment versus treatment using MIPD within the first three days of treatment. | two years
  The percentage of patients with a vancomycin concentration within the therapeutic range (20-25 mg/L) in the first three days after start of treatment for standard of care (flat dose adjusted for renal function) versus MIPD dosing (starting dose determined using pharmacokinetic models).